CLINICAL TRIAL: NCT05419050
Title: A Phase 2 Study of Denosumab for Prevention of Skeletal Disease Progression in Children With Fibrous Dysplasia
Brief Title: Study of Denosumab for Prevention of Skeletal Disease Progression in Children With Fibrous Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000780; 000780-D
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Fibrous Dysplasia
Keywords: McCune-Albright Syndrome
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic | interventions — Denosumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): treatment arm
  Interventions: Drug: denosumab

INTERVENTIONS:
Drug: denosumab — monoclonal antibody to receptor activator of nuclear kappa-B ligand (RANKL), a protein involved in regulating osteoclastogenesis

SUMMARY:
Background:

Fibrous dysplasia (FD) is a disease that affects the bones. It causes bone lesions that can become weak and lead to fractures, deformity, and nerve injuries. FD bone lesions begin to develop soon after birth and grow during childhood. The lesions stop growing in adults but can still cause disability. Researchers want to find ways to stop the growth of FD bone lesions.

Objective:

To test a study drug (denosumab) in children with FD.

Eligibility:

Children aged 4 to 14 years with FD and who are also enrolled in the Screening and Natural History protocol (98-D-0145).

Design:

Participants will have a screening visit at the NIH clinic or by telehealth. Their medical history will be reviewed.

Participants will stay overnight in the hospital 4 times in 76 weeks. Each stay will last 5 to 7 nights.

Participants will also visit a local lab for blood and urine tests every 4 weeks during the study.

Participants will receive denosumab once every 4 weeks for 48 weeks. The medication is given as a shot injected under the skin using a small needle. Some injections may be performed at home by a caregiver. The caregiver will receive training for this procedure.

Participants will undergo many tests that may be repeated throughout the study. They will have a dental exam. They will have tests of their strength and ability to move freely. They will have x-rays and other scans to get pictures of their bones.

Participants will be given another medicine that is administered through a needle in the arm over 30 minutes.

DETAILED DESCRIPTION:
Study Description:

This will be a phase 2, open label, single arm study of denosumab treatment to prevent fibrous dysplasia (FD) lesion progression in children.

Objectives:

Primary Objective:

Evaluate the effect of denosumab on FD lesion progression in children.

Secondary Objectives:

* Evaluate the effects of denosumab on FD lesion activity.
* Evaluate the effect of denosumab on strength and mobility.
* Evaluate the effect of denosumab on pain and quality of life.
* Evaluate the safety and tolerability of denosumab in children with FD.

Endpoints:

Primary Endpoint:

Change in Skeletal Burden Score from baseline to 48 weeks

Secondary Endpoints:

* Percent change in serum bone turnover markers from baseline to 48 weeks: Procollagen 1 Intact N-Terminal Propeptide (P1NP, formation marker), C- telopeptides (CTX, resorption marker), osteocalcin, and bone-specific alkaline phosphatase
* Change in 18F-NaF PET/CT total lesion activity from baseline to 48 weeks
* Change in 18F-NaF PET/CT sentinel lesion intensity (SUVmax) from baseline to 48 weeks
* Change in functional parameters from baseline to 48 weeks, including muscle strength, range-of-motion, and walking speed
* Change in patient-reported outcome scales evaluating pain and quality of life from baseline to 48 weeks, including PROMIS Pediatric measures of Pain Intensity, Pain Interference, Mobility, and Fatigue.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Confirmed diagnosis of fibrous dysplasia
* Age 4 to 14 years
* Concurrent enrollment in the companion Screening and Natural History protocol 98-D-0145
* Provision of signed and dated informed consent form
* Stated willingness of guardian/Legally Authorized Representative (LAR) to comply with all study procedures and availability for the duration of the study
* Ability of guardian/LAR to understand and the willingness to sign a written informed consent document
* For females of reproductive potential: agreement to use highly effective contraception for during study participation. Highly effective contraception methods include:

  * Total abstinence. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Combination of the following (a+b or a+c, or b+c):

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
* Minimum body weight of 12 kilograms

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation
* Known allergic reactions to denosumab
* Prior history, or current evidence, of osteomyelitis/osteonecrosis of the jaw
* Planned invasive dental procedure for the course of the study
* Presence of non-healed dental or oral surgery
* Orthopedic procedure performed less than 6-weeks prior to first day of the denosumab administration (Day 0)
* Acute fracture less than 6-weeks prior to first day of the denosumab administration (Day 0)
* Serum calcium or albumin-adjusted serum calcium below the normal range for the NIH laboratory (patients will be eligible for re-screening after a repletion period lasting up to 6 months)
* 25-hydroxyvitamin D level than 20 ng/mL (patients will be eligible for re screening after a repletion period lasting up to 6 months)
* Untreated or inadequately treated hypophosphatemia as determined by the principal investigator (patients will be eligible for re-screening after initiation or optimization of phosphorus replacement no longer than 6 months)
* Inability to comply with a non-sedated 18F-NaF PET/CT (subjects will be eligible for re- screening after 6 months)
* Use of another investigational agent within the last 3 months prior to the first day of the denosumab administration (Day 0)
* Have any condition which in the opinion of the PI could present a concern for subject safety or difficulty with data interpretation.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Skeletal Burden Score | 48 weeks
  Skeletal Burden Score is a validated measure for quantifying FD disease burden shown to correlate with skeletal outcomes

SECONDARY OUTCOMES:
Percent change in serum bone turnover markers from baseline to 48 weeks: procollagen 1 propeptide (P1NP, formation marker), beta crosslaps telopeptides (CTX, resorption marker), osteocalcin, and bone-specific alkaline phosphatase | 48 weeks
  reflect underlying bone turnover, and correlate with skeletal outcomes
Adverse events | 76 weeks
  Safety endpoints for expected and unexpected adverse events
Change in functional parameters: - Muscle strength - Range-of-motion - Walking speed (6-minute walk) | 48 weeks
  Outcome measures that reflect activities of daily living
Change in 18F-NaF PET/CT total lesion activity from baseline to 48 weeks | 48 weeks
  reflect underlying lesion activity and correlate with skeletal outcomes
Change in patient-reported outcome scales: - SF10 - Brief Pain Inventory - Brief Fatigue Inventory | 48 weeks
  Outcome measures to determine pain and quality of life
Change in 18F-NaF PET/CT sentinel lesion intensity (SUVmax) | 48 weeks
  reflect underlying lesion activity and correlate with skeletal outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Boyce, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: Data will be shared on reasonable request to the PI

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000780-D.html